CLINICAL TRIAL: NCT07035314
Title: The Effect of Systemic Nonsteroidal Anti-inflammatory Drugs (NSAIDs) Vs Intraoperative Infiltration of Steroids in Tonsillar Bed Following Tonsillectomy on Post Tonsillectomy Pain: A Prospective Randomized Controlled Study.
Brief Title: The Effect of Systemic Nonsteroidal Anti-inflammatory Drugs (NSAIDs) Vs Intraoperative Infiltration of Steroids in Tonsillar Bed Following Tonsillectomy on Post Tonsillectomy Pain.
Acronym: NSAIDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS 41/2025
Record Dates: First submitted 2025-04-04; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Tonsillitis Chronic; Tonsillitis Recurrent; OSA - Obstructive Sleep Apnea
Keywords: tonsillitis; tonsillectomy; post tonsillectomy pain; Dexamethasone infiltration in tonsillar bed; NSAIDs
MeSH Terms: conditions — Sleep Apnea, Obstructive; Tonsillitis | interventions — Dexamethasone; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Steroids

STUDY DESIGN:
Intervention Model Description: 3 groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1- First group: will receive local infiltration of steroids (dexamethasone) in tonsillar bed and par (Experimental): 1- First group: will receive local infiltration of steroids (dexamethasone) in tonsillar bed and par
  Interventions: Procedure: Dexamethasone
- 2- Second group: will receive systemic nonsteroidal anti-inflammatory drugs in the analgesic and ant (Experimental): 2- Second group: will receive systemic nonsteroidal anti-inflammatory drugs in the analgesic and anti-inflammatory dosage and paracetamol.
  Interventions: Drug: NSAIDs
- 3- Third group: control group will receive NSAIDs, steroids and paracetamol as standard post tonsill (Active Comparator): 3- Third group: control group will receive NSAIDs, steroids and paracetamol as standard post tonsill
  Interventions: Drug: Control (Standard treatment)

INTERVENTIONS:
Procedure: Dexamethasone — 1- First group: will receive local infiltration of steroids (dexamethasone) in tonsillar bed and paracetamol.
  Other Names: 1- First group: will receive local infiltration of steroids (dexamethasone) in tonsillar bed and paracetamol.
  Arms: 1- First group: will receive local infiltration of steroids (dexamethasone) in tonsillar bed and par
Drug: NSAIDs — 2- Second group: will receive systemic nonsteroidal anti-inflammatory drugs in the analgesic and anti-inflammatory dosage and paracetamol.
  Other Names: 2- Second group: will receive systemic nonsteroidal anti-inflammatory drugs in the analgesic and anti-inflammatory dosage and paracetamol.
  Arms: 2- Second group: will receive systemic nonsteroidal anti-inflammatory drugs in the analgesic and ant
Drug: Control (Standard treatment) — 3- Third group: control group will receive NSAIDs, steroids and paracetamol as standard post tonsillectomy medications in our department.
  Other Names: 3- Third group: control group will receive NSAIDs, steroids and paracetamol as standard post tonsillectomy medications in our department.
  Arms: 3- Third group: control group will receive NSAIDs, steroids and paracetamol as standard post tonsill

SUMMARY:
The aim of this study is to compare the efficacy of adding paracetamol to systemic non-steroidal anti-inflammatory drugs (NSAIDs) versus adding dexamethasone as local infiltration to paracetamol on post tonsillectomy pain control.

DETAILED DESCRIPTION:
A Prospective Randomized Controlled study. The study will be conducted at Ain Shams University hospital, Otolaryngology Department. Study period is 6 months from approval of the protocol. Study Participants will be recruited from outpatient ENT clinic, and ENT department inpatients.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 4-10 years.
* Indications of tonsillectomy such as:

  * Recurrent acute attacks at least 7 episodes in the past year or at least 5 episodes per year for 2 years or at least 3 episodes per year for 3 years.
  * Chronic tonsillitis and hypertrophy of tonsils causing sleep apnea, difficulty in deglutition, interference in speech.
* Tonsillectomy by cold dissection only.
* American Society of Anesthesiologists (ASA) classification 1,2 (Normal Health, Mild systematic disease).

Exclusion Criteria:

* Patients with age less than 4 and more than 10 years.
* Indications of tonsillectomy other than chronic tonsillitis such as lymphoma.
* Patients on chronic steroid therapy
* Hemoglobin level less than 10 gm/dL
* Presence of acute infection in the upper respiratory tract, acute tonsillitis
* American Society of Anesthesiologists (ASA) classification ASA 3,4 (Severe systematic disease such as uncontrolled Diabetes, cardiac disease, liver or kidney disease, life threating medical conditions)
* Regular use of analgesics within a week of surgery.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
post tonsillectomy pain | DAY 0 6h, 24h post-operatively and DAY 5 post-operatively
  The primary endpoints that will be used is resting pain scores using virtual analogue scale; VAS score (0: no pain-10: worst pain) at DAY 0 after 6h, 24h and DAY 5 post-operatively. Where pain score will be measured at multiple points during the outcome intervals, the pain scores at the time closest to six and 24h will be used.

SECONDARY OUTCOMES:
Additional pain medication needed | 2 weeks post operatively
  The percentage of the patients in group 1 and 2 that will need extra analgesia
Pt feedback after tonsillectomy | 2 weeks post operatively
  Patient satisfaction and return to normal activity.
Complications | 2 weeks post operatively
  Adverse effects noticed such as nausea, vomiting, infection and post tonsillectomy bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verma RR, Sriraman R, Rana SK, Ponnanna NM, Rajendar B, Ghantasala P, Rajendra L, Matur RV, Srinivasan VA. E6 protein of human papillomavirus 16 (HPV16) expressed in Escherichia coli sans a stretch of hydrophobic amino acids, enables purification of GST-DeltaE6 in the soluble form and retains the binding ability to p53. Protein Expr Purif. 2013 Nov;92(1):41-7. doi: 10.1016/j.pep.2013.08.010. Epub 2013 Sep 6. PMID 24012792

DOCUMENTS (1):
  • Study Protocol (2025-01-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT07035314/Prot_000.pdf